CLINICAL TRIAL: NCT01405066
Title: CT Technologists Dose Audit Reports and Educational Seminar to Reduce Patient Radiation Exposure From Medical Imaging
Brief Title: Radiation Dose Audit Reports to Reduce Radiation Exposure From CT Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GroupHealthCoop Foundation2011
Record Dates: First submitted 2011-07-21; First posted 2011-07-29 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Decrease Variability and Amount of Radiation Dose From CT Exams
Keywords: Computed Tomography (CT); Ionizing radiation; Advanced medical imaging; Radiation Dose Audit Reports

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Reports and Educational Seminar (Experimental)
  Interventions: Behavioral: Radiation Dose Audit Reports; Behavioral: Educational Seminar: Radiation Dose Reduction

INTERVENTIONS:
Behavioral: Radiation Dose Audit Reports — Audit reports by CT technologist, with graphs of radiation dose levels of 20 exams from each of the 4 most common CT exams. Reports show the distribution of radiation dose levels by each exam type, and compares the technologist's dose levels to the overall levels from the clinic where they work and to the United Kingdom's 2003 Reference Dose. Prior to the graphs, the reports include an introductory page explaining the organization of the report and defining the dosimetry metrics. The final page of the report lists exams meriting individual review because their doses are higher than that of the clinic averages.
Behavioral: Educational Seminar: Radiation Dose Reduction — Seminar led by a Radiologic Physicist and Radiologist. Discussion of the parameters associated with radiation dosage from CT exams and methods for changing these parameters to lower radiation dose.

SUMMARY:
The purpose of this study is to quantify variation in radiation dose levels across CT technologists, and determine the effectiveness of combining radiation dose audit reports and an educational seminar as a means to reduce the variation and level of patient exposure to radiation.

The investigators expect the radiation dose audit reports and educational seminar will lead to reduced radiation exposure to patients by making technologists more aware of the risks of radiation exposure from CT exams and identifying technologists with higher radiation exams compared with their peers.

The investigators expect the degree to which a technologist is concerned and aware about radiation exposure and cancer risk will be associated with adherence to radiation reduction protocols and the subsequent level of radiation their patients are exposed to when receiving a CT examination.

DETAILED DESCRIPTION:
The use of advanced diagnostic imaging has increased dramatically over the past decade, not only contributing to rising medical costs but also exposure to ionizing radiation, of which CT imaging plays a prominent role because it requires a relatively high dose of radiation to produce an image when compared to conventional X-rays. The growth in the use of CT imaging along with all other advanced medical imaging has been well documented, and taken as a whole the use of these services has grown quicker than all other services provided by physicians. Research has also shown great variability in the amount of radiation exposure to individual patients, even when patient and other characteristics are controlled for. Given the increase in the use of CT imaging and the variability in radiation exposure between similar imaging exams, it is important to study ways of standardizing and reducing radiation levels from CT imaging. Little is understood about the role of CT technologists' attitudes and how they may influence patient radiation exposure, therefore, this project also give us the opportunity to survey the technologists and determine if there is a relationship between technologist attitudes and awareness and the radiation exposure of patients.

ELIGIBILITY:
Inclusion Criteria:

* Group Health CT Technologist from Capitol Hill, Tacoma and Bellevue Clinics

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Radiation dose levels (measured by dose linear product (DLP) and effective dose (ED)) from CT exams as a measure of the effectiveness of radiation dose audit reporting and educational intervention for lowering patient exposure to radiation from CT exams. | April 2011 and September 2011
  We will report dose data at two time points, April 2011 (data for these reports collect from November 2010 to March 2011), and September 2011 (data collected from April 2011 to August 2011), and compare the data from the two time points to see if there was a change in dose levels (DLP and ED) for the time period (April to August) after the presentation of the first audit reports and delivery of the educational interventions to the CT technologists.

SECONDARY OUTCOMES:
CT Tech technologists attitudes and awareness towards radiation exposure from CT imaging | April 2011 to September 2011

CONTACTS AND LOCATIONS:
Overall Officials: Diana Miglioretti, PhD, Principal Investigator — Group Health Research Institute